CLINICAL TRIAL: NCT06581939
Title: Impact of an Early and Extended Rehabilitation Program Combining Individually Tailored Nutrition and Physical Activities on Patient Outcomes After Invasive Mechanical Ventilation and Vasopressor Therapy in the ICU : A Multicenter Randomized Controlled Trial
Brief Title: Impact of an Early and Extended Rehabilitation Program Combining Individually Tailored Nutrition and Physical Activities on Patient Outcomes After Invasive Mechanical Ventilation and Vasopressor Therapy in the ICU
Acronym: NUTRIREA-4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC23_0585
Record Dates: First submitted 2024-08-20; First posted 2024-09-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mechanical Ventilation
Keywords: Critical care; Nutritional support; Mechanical ventilation; Shock; Macronutrients; Rehabilitation; Physiotherapy; Adapted physical activity
MeSH Terms: conditions — Shock | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental): Individualized rehabilitation program
  Interventions: Procedure: Rehabilitation group
- Control group (Active Comparator): Usual care
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Rehabilitation group — In the rehabilitation group, patients will follow an individualized rehabilitation program started early in the ICU and continued in the post-ICU ward then at home for 12 weeks, combining goal-directed nutrition and physical activity, tailored to gains made over time by each patient, with the involvement of dieticians, physiotherapists, and adapted-physical-activity instructors.
  Arms: Rehabilitation group
Procedure: Control group — In the control group, patients will receive usual care from day-0 to day-180.
  Arms: Control group

SUMMARY:
The NUTRIREA-4 trial will test the hypothesis that an individually tailored rehabilitation program combining nutritional therapy, physiotherapy, and physical activity and started early in the ICU then continued uninterruptedly throughout the post-ICU stay and at home after hospital discharge improves the long-term outcomes of critical-illness survivors, compared to usual care.

From ICU admission to recovery at home, the trial patients will receive either usual care or the early extended rehabilitation program. Usual care will consist in nutritional support and physiotherapy according to usual local practice in each participating ICU. The early extended program will consist of nutritional therapy, physiotherapy, and physical activity according to a standardized protocol tailored to general- and muscle-health improvements achieved in each individual patient over time.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation (MV) started in the ICU within the past 24 h, or started before ICU admission with ICU admission within the past 24 h, and expected to be required for at least 48 hours after randomization
* Treatment with a vasoactive agent for shock (adrenaline, dobutamine, or noradrenaline)
* Nutritional support expected to be started within 24 h after intubation (or within 24 h after ICU admission if intubation occurred before ICU admission)
* Age 18 or older
* Patient and/or next-of-kin informed about the trial and having consented to participation in the trial. If the patient is unable to receive information and no next-of-kin can be contacted during screening for the trial, trial inclusion will be completed as an emergency procedure by the ICU physician, in compliance with French law.
* Covered by the French public health-insurance system

Exclusion Criteria:

* MV started more than 24 hours earlier
* Specific nutritional needs, such as pre-existing long-term home enteral or parenteral nutrition for chronic bowel disease
* Dying patient, do-not-resuscitate order, or other treatment- limitation decision at ICU admission
* Social circumstances hindering follow-up and telephone/video consultations (no fixed address, non-European residence)
* Inability to provide a stable personal mobile phone number (temporary number or not in the owner's name)
* Communication difficulties via telephone or video consultation (pre-existing severe hearing or visual impairment)
* Pre-existing chronic illness with life expectancy <6 months
* Pre-existing cognitive impairment
* Pre-existing spinal injury
* Inability to walk before the critical illness
* Acute or chronic neuromuscular disease
* Brain injury, e.g., due to cardiac arrest, stroke, or severe trauma
* Pregnancy, recent delivery, or lactation
* Adult under guardianship
* Correctional facility inmate
* Institutionalized patient
* Prior inclusion in a randomized trial designed to compare rehabilitation programs delivered to patients during critical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
6-minute-walk distance | 6 months
  The primary endpoint is the 6-minute-walk distance (6MWD), in meters, assessed by blinded physicians and research nurses during a hospital visit 6 months after randomization.

SECONDARY OUTCOMES:
Handgrip strength | 6 months after randomization
  Handgrip strength (Kg and percent of predicted strength) at 6 months after randomization
Medical Research Council (MRC) score | 6 months after randomization
  MRC score at 6 months after randomization
Muscle mass assessed by the mid-arm muscle circumference (MAMC) | 6 months after randomization
  MAMC at 6 months after randomization
Physical activity assessed by the International Physical Activity Questionnaire Short Form (IPAQ-SF) | 3 months after randomization
  IPAQ-SF score at 3 months after randomization
Physical activity assessed by the International Physical Activity Questionnaire Short Form (IPAQ-SF) | 4 months after randomization
  IPAQ-SF score at 4 months after randomization
Physical activity assessed by the International Physical Activity Questionnaire Short Form (IPAQ-SF) | 5 months after randomization
  IPAQ-SF score at 5 months after randomization
Physical activity assessed by the International Physical Activity Questionnaire Short Form (IPAQ-SF) | 6 months after randomization
  IPAQ-SF score at 6 months after randomization
Physical activity assessed by the International Physical Activity Questionnaire Short Form (IPAQ-SF) | 12 months after randomization
  IPAQ-SF score at 12 months after randomization
Calorie intakes | From day 0 to 12 months
  Calorie intakes (daily mean during the hospital stay and at home at D90, D120, D150, D180, and one year after randomization)
Protein intakes | From day 0 to 12 months
  Protein intakes (daily mean during the hospital stay and at home at D90, D120, D150, D180, and one year after randomization)
Body weight | 6 months
  Mean changes in body weight measured at 6 months)
Mortality rates | Day 90
  90-day mortality rates
Mortality rates | 6 months
  6-month mortality rates
Mortality rates | 12 months
  12-months mortality rates
Hypoglycemia | From day 0 to day 7
  Proportion of patients with at least one hypoglycemia from day 0 to day 7
Blood glucose | From day 0 to day 7
  Mean blood glucose from day 0 to day 7
Quality of life assessed using the Short Form 36 Health Survey (SF-36) | 6 and 12 months
  SF-36 scores 6 and 12 months after randomization
Handgrip strength | ICU discharge, an average of 10 days
  Handgrip strength (Kg and percent of predicted strength) at ICU discharge
Handgrip strength | Hospital discharge, an average of 20 days
  Handgrip strength (Kg and percent of predicted strength) at hospital discharge
Medical Research Council (MRC) score | ICU discharge, an average of 10 days
  MRC score at ICU discharge
Medical Research Council (MRC) score | Hospital discharge, an average of 20 days
  MRC score at hospital discharge
Muscle mass assessed by the mid-arm muscle circumference (MAMC) | ICU discharge, an average of 10 days
  MAMC at ICU discharge
Muscle mass assessed by the mid-arm muscle circumference (MAMC) | Hospital discharge, an average of 20 days
  MAMC at hospital discharge
Body weight | ICU discharge, an average of 10 days
  Mean changes in body weight measured at ICU discharge
Mortality rates | ICU discharge, an average of 10 days
  ICU discharge mortality rates
Mechanical Ventilation (MV) duration | From D0 until the date of cessation of mechanical ventilation, an average of 7 days
  Days of MV
ICU-acquired infection | From day 0 until the date of discharge from ICU, an average of 10 days
  Proportion of patients with at least one ICU-acquired infection
ICU and hospital stay lengths | From day 0 until the day of discharge from hospital, an average of 20 days
  ICU and hospital stay lengths (days)
Mortality rates | Hospital discharge, an average of 20 days
  Hospital discharge mortality rates
Insulin | From day 0 until the date of ICU discharge, an average of 10 days
  Days on insulin in the ICU
Delay from randomization to first standing-up | From date of randomization until the date of first standing-up, an average of 7 days
  Delay from randomization to first standing-up (days)
Delay from randomization to first walking | From date of randomization until the date of first walking, an average of 15 days
  Delay from randomization to first walking (days)

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 6 and 12 months
  HADS score 6 and 12 months after randomization
Post-traumatic stress disorder Check List for DSM-5 (PCL-5) | 6 and 12 months
  PCL-5 score 6 and 12 months after randomization
Resilience assessed using the Connor-Davidson Resilience Scale (CD-RISC10) | 6 and 12 months
  CD-RISC-10 6 and 12 months after randomization
Posttraumatic growth using the Posttraumatic Growth Inventory Short Form (PTGI-SF) | 6 and 12 months
  PTGI-SF 6 and 12 months after randomization
Cognitive performance using the Montreal Cognitive Assessment (MoCA) | 6 and 12 months
  MoCA 6 and 12 months after randomization
Qualitative assessment on how the rehabilitation program influences resilience and psychological recovery after ICU | 12 months
  Semi-structured interviews
Time course of circulating Growth-differentiation factor-15 (GDF-15) | Inclusion, H24, H72, Day 7, ICU discharge, Day 180
  GDF-15 plasma level
Effects of the individualized rehabilitation program, compared to usual care, on IFN-γ | Inclusion, H24, H72, Day7, ICU discharge, Day 180
  IFN-γ plasma level
Effects of the individualized rehabilitation program, compared to usual care, on IFN-γ | Inclusion, H24, H72, Day7, ICU discharge, Day 180.
  IL-1β plasma level
Effects of the individualized rehabilitation program, compared to usual care, on IL-6 | Inclusion, H24, H72, Day7, ICU discharge, Day 180
  IL-6 plasma level
Effects of the individualized rehabilitation program, compared to usual care, on TNF-α | Inclusion, H24, H72, Day7, ICU discharge, Day 180
  TNF-α plasma level
Effects of the individualized rehabilitation program, compared to usual care, on FGF-21 | Inclusion, H24, H72, Day7, ICU discharge, Day 180
  FGF-21 plasma level
Effects of the individualized rehabilitation program, compared to usual care, on leptin | Inclusion, H24, H72, Day7, ICU discharge, Day 180
  leptin plasma level
Effects of the individualized rehabilitation program, compared to usual care, on C-peptide | inclusion, H24, H72, Day7, ICU discharge, Day 180
  C-peptide plasma level
Effects of the individualized rehabilitation program, compared to usual care, on Ghrelin | Inclusion, H24, H72, Day7, ICU discharge, Day 180
  Ghrelin plasma level

CONTACTS AND LOCATIONS:
Overall Officials: Jean REIGNIER, MD, PhD, Principal Investigator — Nantes University Hospital
Locations (52):
- France (52):
  - CH d'Albi, Albi
  - CHU d'Amiens - Site Sud, Amiens
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH d'Angoulème, Angoulême
  - CH d'Argenteuil, Argenteuil
  - CH de Belfort, Belfort
  - CHU de Besançon, Besançon
  - CH de Béthune, Béthune
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH de Cholet, Cholet
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CH de Dieppe, Dieppe
  - CHU de Dijon, Dijon
  - CH d'Annecy Genevois, Épagny
  - Centre Hospitalier Sud Essonne, Étampes
  - Hôpital Raymond Poincaré - AP-HP, Garches
  - CHU de Grenoble, Grenoble
  - CH d'Haguenau, Haguenau
  - CH de Vendée, La Roche-sur-Yon
  - Hôpital de Bicêtre - AP-HP, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - CH de Lens, Lens
  - CHRU de Lille, Lille
  - CH de Lomme, Lomme
  - CH de Lorient, Lorient
  - CHU de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice - Hôpital Pasteur, Nice
  - CHU de Nice, Nice
  - CH d'Orléans, Orléans
  - Hôpital Saint-Louis - AP-HP, Paris
  - Hôpital Cochin - AP-HP, Paris
  - Hôpital la Pitié-Salpétrière - AP-HP, Paris
  - Hôpital Tenon - AP-HP, Paris
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CH de Saint-Brieuc, Saint-Brieuc
  - Hôpital Delafontaine, Saint-Denis
  - Centre Hospitalier de Saint-Nazaire, Saint-Nazaire
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - CH de Saint-Malo, St-Malo
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU de Tours, Tours
  - CH de Valenciennes, Valenciennes
  - CH de Vannes, Vannes
  - CH de Verdun, Verdun